CLINICAL TRIAL: NCT02511171
Title: A Study to Explore the Acceptability of Parental Blinding in Clinical Trials of Osteopathy With Excessively Crying Infants as Study Participants
Brief Title: Parental Blinding in Clinical Trials of Osteopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European School of Osteopathy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESO-002-Pilot1
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- No intervention (No Intervention): Subjects do not receive osteopathic care
- Cranial osteopathic manipulative treatment (Experimental): Subjects receive individualised osteopathic treatment
  Interventions: Other: Cranial osteopathic manipulative therapy

INTERVENTIONS:
Other: Cranial osteopathic manipulative therapy
  Other Names: Cranial osteopathy
  Arms: Cranial osteopathic manipulative treatment

SUMMARY:
The aim of this research is to assess the acceptability of using a mobile folding screen for blinding parents of infant study participants in clinical trials of osteopathic interventions. The preliminary data of this acceptability study will inform future randomized controlled trials with infant participants where parental blinding is required. 30 excessively crying infants will be randomly allocated to 2 groups, one group receives osteopathic intervention, the other group does not receive treatment. All infants are treated (or not) behind a mobile folding screen, so that parents are not aware of group allocation. After a 'treatment' period of 20 min, the screen is removed, and parents are asked to fill in an acceptability and blinding success questionnaire.

DETAILED DESCRIPTION:
Parents who take part in the research will arrive at their scheduled appointment. If parents have not brought their signed consent form, they will be asked to sign it in clinic. This consent form also will contain questions about infant and parent demographics as well as socio-demographic background details, which the parent is asked to fill in. Parents will be guided into a separate treatment room, which contains a treatment table behind a screen. A qualified osteopathic practitioner will take the case history for each infant who then receives a physical assessment. After that, the parent will have to give consent for the infant to be further involved in the study and to be treated. This procedure will be done without the screen, so that the parent can see what is going on. Then the infant is placed behind the screen on the treatment couch. The osteopath will be informed by the Research Assistant whether the infant is allocated (via random allocation list) to receiving either no intervention or OMT for 20 min. For infants in the OMT group, the osteopathic practitioner will carry out the treatment procedure, and the Research Assistant will act as an intermediary. Infants in the 'no intervention' group will just lie on the couch, without being touched by the osteopath.

At all times, the screen is placed between the parent and their infant on the treatment couch, so that the parent will not be able to see their infant. However, the intermediary is placed in a way so that the parent can see and communicate with them, and the intermediary can observe what is happening behind the screen with the infant. The osteopathic practitioner will be present at all times in both groups, to safeguard the infant from rolling off the couch in case the infant does not receive any intervention. In addition, if the infant starts crying, the osteopathic practitioner will try to calm the infant down (for infants in the OMT group the osteopath will use toys and touch, in the 'no intervention' group toys only will be used, no touch), but if necessary will ask the parent to come round the screen and help in calming their infant down. If this is the case, the osteopathic practitioner stops the treatment, if the infant is placed in the OMT group, and waits until the infant is calmed down so that the parent can go back behind the screen. This procedure will be repeated until 20 min of the treatment period are over. The same procedure applies for the 'no intervention group', except that the osteopath will not touch the infant, rather tries to calm it down with toys or eventually will call the parent in to do the calming. After the 20mins of 'treatment period', parents of infants in both groups are required to fill in the blinding success and acceptability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged up to four months, crying for more than three hours per day, some of the crying is in-consolable; parents have signed a consent form to take part in the study

Exclusion Criteria:

* Infants who are not safe to treat as a result of the osteopathic assessment procedure, infants where no inconsolable crying is reported by parent

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blinding success and acceptability questionnaire (non-validated) | up to 5 min
  Parents are asked whether they found aspects of the treatment environment (intermediary, screen) acceptable or not, they are also asked which group they believed their child was placed in

CONTACTS AND LOCATIONS:
Locations (1):
- European School of Osteopathy, Maidstone, Kent, United Kingdom

REFERENCES:
- [Background] Miller JE, Newell D, Bolton JE. Efficacy of chiropractic manual therapy on infant colic: a pragmatic single-blind, randomized controlled trial. J Manipulative Physiol Ther. 2012 Oct;35(8):600-7. doi: 10.1016/j.jmpt.2012.09.010. PMID 23158465